CLINICAL TRIAL: NCT02499562
Title: Randomed and Double-blinded Phase II Clinical Trial of Hydronidone Capsules(F351) in Patients With Liver Fibrosis Induced by HBV Chronic Hepatitis
Brief Title: A Phase II Clinical Trial of Hydronidone Capsules(F351) in Patients With Liver Fibrosis Induced by HBV Chronic Hepatitis
Acronym: HBV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Genomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNI-F351-201402
Record Dates: First submitted 2015-06-26; First posted 2015-07-16 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — hydronidone; 5-methyl-1-(4-hydroxylphenyl)-2-(1H)-pyridone; entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hydronidone(180mg) & Entecavir & Placebo (Experimental): hydronidone capsule 30mg/capsule hydronidone capsule, three times a day, 2 capsules each time; with co-administration of placebo capsule, three times a day, 2 capsules each time, namely the daily dose of the investigational product is 180mg.
  The test groups and the control group take the entecavir capsule which is orally taken for antiviral therapy, one time a day, 0.5mg each time, oral administration on an empty stomach.
  Interventions: Drug: Hydronidone; Drug: Placebo; Drug: Entecavir
- Hydronidone(270mg) & Entecavir & Placebo (Experimental): hydronidone capsule 30mg/capsule hydronidone capsule, three times a day, 3 capsules each time; with co-administration of placebo capsule, three times a day, 1 capsules each time, namely the daily dose of the investigational product is 270mg.
  The test groups and the control group take the entecavir capsule which is orally taken for antiviral therapy, one time a day, 0.5mg each time, oral administration on an empty stomach.
  Interventions: Drug: Hydronidone; Drug: Placebo; Drug: Entecavir
- Hydronidone(360mg) & Entecavir (Experimental): hydronidone capsule 30mg/capsule hydronidone capsule, three times a day, 4 capsules each time; namely the daily dose of the investigational product is 360mg.
  The test groups and the control group take the entecavir capsule which is orally taken for antiviral therapy, one time a day, 0.5mg each time, oral administration on an empty stomach.
  Interventions: Drug: Hydronidone; Drug: Entecavir
- Entecavir & Placebo(360mg) (Experimental): placebo capsule 30mg/capsule placebo capsule, three times a day, 4 capsules each time. The test groups and the control group take the entecavir capsule which is orally taken for antiviral therapy, one time a day, 0.5mg each time, oral administration on an empty stomach.
  Interventions: Drug: Placebo; Drug: Entecavir

INTERVENTIONS:
Drug: Hydronidone — The investigational products in the test groups and control group shall be orally taken 30 minutes before meals for 52 continuous weeks. There are respectively 60 cases in the test group I, II, III and the control group, totally 240 cases.
  Other Names: F351
  Arms: Hydronidone(180mg) & Entecavir & Placebo; Hydronidone(270mg) & Entecavir & Placebo; Hydronidone(360mg) & Entecavir
Drug: Placebo
  Arms: Entecavir & Placebo(360mg); Hydronidone(180mg) & Entecavir & Placebo; Hydronidone(270mg) & Entecavir & Placebo
Drug: Entecavir

SUMMARY:
To explore the effective dose and safety of the effect of hydronidone and entecavir on hepatic fibrosis in chronic viral hepatitis B.

DETAILED DESCRIPTION:
Primary observation indexes:

Hepatic fibrosis Ishak score after treatment decreases by the proportion not less than 1 compared with that before treatment.

Secondary observation indexes :

1. Negative conversion ratio of HBV DNA after treatment (HBV DNA<1×103copies/mL) and falling range.
2. The falling proportion of Fibrocan Kpa value after treatment compared with that before treatment.
3. The falling proportion that decreases not less than 1 level and progression-free fibrosis after treatment compared with that before treatment.
4. The improvement of ALT of liver function.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65, all genders.
2. History of chronic hepatitis B, HBsAg positive≧six months.
3. ALT<eight-fold ULN (maximum).
4. Significant liver fibrosis confirmed by liver biopsy.
5. HBeAg positive patients, HBV DNA>2.0×104 IU/mL (copies/mL); HBeAg negative patients，HBV DNA>2.0×103 IU/mL (104copies/mL).
6. Having not accepted the antiviral therapy with interferon and/or nucleoside analog.
7. Having not taken anti-inflammatory drugs to protect liver within 1 month before selection.
8. Capable of understanding and signing the informed consent before the study.

Exclusion Criteria:

1. Failing to meet any one requirement of the inclusion criteria.
2. Having suffered massive hemorrhage of gastrointestinal tract within 3 months before selection
3. TBiL>three-fold ULN.
4. AFP>100 ug/L
5. PLT≦60×109/L
6. PTA<50%
7. Having obvious space-occupying lesion in liver as shown by B ultrasound examination.
8. With a portal vein ≧1.2cm wide as shown by B ultrasound examination.
9. BMI index>30.
10. The patient who suffered from liver function decompensation hepatic cirrhosis and liver neoplasms.
11. The patient with alcoholic, drug-induced, hereditary, immune and other viral and non- viral chronic hepatitis.
12. The patient with angiocarpy, lung, kidney, incretion, nerve and blood system disease and mental disease.
13. The patient with active peptic ulcer.
14. Gestational and breast feeding women.
15. The subject is the legal disabled person according to the Law of the People's Republic of China on the Protection of Disabled Persons of the April 2008 edition.
16. The subject who participated in other drug tests within recent 3 months.
17. The patient who is suspected with poor compliance or disagrees to participate in the test.
18. The patient who is considered by other investigators not to be suitable for participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-06-25; Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Changes in hepatic fibrosis in chronic viral hepatitis B | one year

CONTACTS AND LOCATIONS:
Overall Officials: LunGen Lu, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Jun Cheng, Principal Investigator — Beijing Ditan Hospital
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Beijing

REFERENCES:
- [Derived] Cai X, Liu X, Xie W, Ma A, Tan Y, Shang J, Zhang J, Chen C, Yu Y, Qu Y, Zhang L, Luo Y, Yin P, Cheng J, Lu L. Hydronidone for the Treatment of Liver Fibrosis Related to Chronic Hepatitis B: A Phase 2 Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1893-1901.e7. doi: 10.1016/j.cgh.2022.05.056. Epub 2022 Jul 13. PMID 35842120